CLINICAL TRIAL: NCT06736886
Title: Effect of Light Color Temperature Applied During Breastfeeding on Mother's Stress, Anxiety, Peace and Breastfeeding Motivation: A Randomized Controlled Trial
Brief Title: Effect of Light Color Temperature Applied During Breastfeeding on Mother's Stress, Anxiety, Peace and Breastfeeding Motivation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Emine Yıldırım, Assistant professor, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2053231
Record Dates: First submitted 2024-12-05; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Light; Stress; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Light application
  Interventions: Other: Light application
- control group (Placebo Comparator): Light application
  Interventions: Other: Light application

INTERVENTIONS:
Other: Light application — Light application

SUMMARY:
Breastfeeding is an important condition for the health of the mother and the baby, which is the most difficult for mothers after birth. Since it is an important practice for both the mother and the baby, the evaluation and reduction of the mother's stress factors can help the hospital to regulate the lighting of the breastfeeding room. In addition, setting the light color temperature to a more appropriate kelvin can make a positive contribution to the hospital in terms of costs. For this purpose, when researchers look at the literature, we have not come across a randomized controlled study examining the effect of the light color temperature applied during breastfeeding on the mother's stress, anxiety, peace and breastfeeding motivation. Researchers' purpose is to determine the effect of the light color temperature applied during breastfeeding on the mother's stress, anxiety, peace and breastfeeding motivation.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have given birth for the first time,
* being 18 years of age and older,
* volunteering.

Exclusion Criteria:

* Being a mother who has given birth to more than one child,
* having any problem that prevents communication (such as not knowing Turkish, having hearing, speaking and understanding disorders),
* receiving psychiatric treatment (pharmacotherapy or psychotherapy),
* having a disease that prevents vision.

Ages: 18 Hours to 45 Hours | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
stress scale | 2 minutes
  QUESTIONNAIRE
anxiety scale | 2 minutes
  QUESTIONNAIRE

IPD SHARING:
Plan to Share IPD: No
Can be shared when necessary